CLINICAL TRIAL: NCT04258878
Title: Prospective Cohort Study in Evaluation of Risk Factors for Infection During and After Coronary Graft Operations.
Status: Unknown | Type: Observational
Last Known Status: Not yet recruiting
Sponsor: Assiut University (Other)
Responsible Party: Principal Investigator, Mohammed Hussein Rushdi, Dr, Assiut University
Other Study IDs: periop- RFs in cardiac surgery
Record Dates: First submitted 2018-09-05; First posted 2020-02-06 (Actual); Last update posted 2020-02-06 (Actual); Status verified 2020-02

CONDITIONS: Surgical Wound Infection
MeSH Terms: conditions — Surgical Wound Infection | interventions — Sternotomy

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 2 Years
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Procedure: Sternotomy — Procedure: Sternotomy for coronary artery bypass graft, valvuloplasty, aortic surgery or combined procedures, under extracorporeal circulation or not, in emergency or scheduled.

SUMMARY:
We aim to prospectively evaluate the risk factors that can play a role before, during or after the surgical period.

DETAILED DESCRIPTION:
Surgical site infections (SSIs) are either superficial or deep and may involve the organs, or spaces accessed during an operation. The reported incidence of SSIs in coronary artery bypass grafting (CABG) surgery ranges between 0.3% and 8%.

There is a strong suggestion that an impairment of vascular supply of the sternum may be one of the most important factors influencing the incidence of deep sternal wound infection (DSWI). Several studies have studied the risk factors for SSIs including DSWI in cardiac surgery. These risk factors included obesity, diabetes mellitus, chronic obstructive pulmonary disease (COPD), connective tissue disease, steroid use, smoking, peripheral vascular disease and renal insufficiency. In addition, intraoperative factors (e.g., use of bilateral internal mammary arteries [BIMA] grafting, prolonged cardiopulmonary bypass [CPB] duration) and postoperative variables (e.g., prolonged mechanical ventilation, reoperation for bleeding, postoperative transfusions and gastrointestinal, nephrological and respiratory complications) have been shown to be associated with DSWI.

The risk for sternal wound infection (SWI) is increased if cardiac surgery involves internal thoracic arteries grafting and a valve procedure, or use of a ventricular assist device.

Leg wound infections at donor sites account for >70% of cases with severe infection following cardiac surgery.

Cardiac SSIs increase the length of hospital stay (LOS) and increase treatment costs in proportion to the severity of the infection. These costs increase by 3.8%, 14.7% and 29.4% in mild, moderate and severe infections respectively.

Treatment is often confounded by the emergence of antibiotic-resistant pathogens and in addition, substantial proportions of these infected patients are elderly and have co-existing medical problems. In the past, such elderly patients with significant comorbidities would not have been considered for surgery.[8] As the population ages, it is reasonable to assume that older and sicker patients will be admitted for surgery, and this will inevitably increase the risk and incidence of SSIs.

ELIGIBILITY:
IInclusion Criteria:

1. patient aged more than 18 yards old
2. sternotomy for: coronary artery bypass,

Exclusion Criteria:

1. patient under age or 18years old.
2. patient who has endocarditis.
3. patient who underwent surgery with prothetic material, within the 12 months preceeding cardiac procedure.

Ages: 18 Years to 70 Years | Sex: All
Age Groups: Adult, Older Adult
Study Population: All patients who presented to Cardiothoracic Surgery Department, Assiut University Heart Hospital who will undergo coronary artery bypass surgery.
Sampling Method: Probability Sample
Enrollment: 100 (Estimated)
Dates: Start 2020-04-01 (Estimated); Primary Completion 2021-03-29 (Estimated); Study Completion 2022-04-30 (Estimated)

PRIMARY OUTCOMES:
surgical wound infection | baseline
  Evaluate the duration of complete healing of the sternum :By
  1. Radiological (chest x-ray ant-post view and lat view in first 3 weeks post-operative
  2. Clinical examination in first 3 weeks post operative

SECONDARY OUTCOMES:
Evaluation of perioperative risk factors for surgical wound infection in cardiac surgery | baseline
  1. Evaluate rate of wound infection in first 3 weeks post operative
  2. -Evaluate the improvement in symptoms of patients postoperative: By
     1. pain by pain score in first 3 week post operative
     2. regain normal activity in first 3 week post operative

CONTACTS AND LOCATIONS:
Overall Officials: Mahmoud Khairy El-Haish, Prof, Study Director — Assuit University Hospital